CLINICAL TRIAL: NCT06874725
Title: Directly Observed Preventive Therapy (DOPT) for Latent Tuberculosis Infection Patients With Poorly Controlled Diabetes Mellitus
Brief Title: Latent Tuberculosis in Type 2 Diabetes
Acronym: TB
Status: Active, not recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Taichung Veterans General Hospital (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: TCVGH-CE18090B
Record Dates: First submitted 2025-03-08; First posted 2025-03-13 (Actual); Last update posted 2025-03-13 (Actual); Status verified 2025-03

CONDITIONS: Latent Tuberculosis Infection
Keywords: Latent tuberculosis infection; diabetes; observational study
MeSH Terms: conditions — Latent Tuberculosis; Diabetes Mellitus | interventions — rifapentine; Isoniazid

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- 3 months of weekly rifapentine plus isoniazid (Active Comparator): 3 months of weekly rifapentine plus isoniazid
  Interventions: Drug: Rifapentine and Isoniazid for 3 months
- 9 months of daily isoniazid (Active Comparator): 9 months of daily isoniazid
  Interventions: Drug: Isoniazid (INH) daily for 9 months

INTERVENTIONS:
Drug: Rifapentine and Isoniazid for 3 months — tuberculosis preventive therapy (TPT) with 3 months of weekly rifapentine plus isoniazid (3HP)
  Other Names: 3HP
  Arms: 3 months of weekly rifapentine plus isoniazid
Drug: Isoniazid (INH) daily for 9 months — tuberculosis preventive therapy (TPT) with 9 months of daily isoniazid (9H)
  Other Names: 9H
  Arms: 9 months of daily isoniazid

SUMMARY:
The patients with poorly controlled DM underwent LTBI screening by using QuantiFERON (QFT). QFT-positivity predictors were evaluated. The patients with LTBI received tuberculosis preventive therapy, 9 months of daily isoniazid (9H) or 3 months of weekly rifapentine plus isoniazid (3HP), administered by pulmonologists. The completion rates and inflammatory markers were also investigated.

DETAILED DESCRIPTION:
Poor control of diabetes mellitus (DM) increases active tuberculosis (TB) risk. Understanding risk factors for latent TB infection (LTBI) in this population is crucial for policy making. Under a collaborative multidisciplinary team consisting of endocrinologists and pulmonologists, patients with poorly controlled DM were enrolled; these patients underwent LTBI screening by using QuantiFERON (QFT). QFT-positivity predictors were evaluated. The patients with LTBI received tuberculosis preventive therapy, 9 months of daily isoniazid (9H) or 3 months of weekly rifapentine plus isoniazid (3HP), administered by pulmonologists. The completion rates and inflammatory markers were also investigated.

ELIGIBILITY:
Inclusion Criteria:

* aged ≥45 years
* poorly controlled DM (pDM), defined as HbA1c ≥9% within the preceding year

Exclusion Criteria:

* active TB
* immunocompromise (use of immunosuppressors
* current pregnancy

Min Age: 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 552 (Actual)
Dates: Start 2018-04-18 (Actual); Primary Completion 2024-04-30 (Actual); Study Completion 2025-04-18 (Estimated)

PRIMARY OUTCOMES:
Brain-Derived Neurotrophic Factor | 9 months
  Biomarker

SECONDARY OUTCOMES:
Inflammatory markers | 9 months
  aryl hydrocarbon receptor, adhesion molecules, dickkopf-related protein 1

CONTACTS AND LOCATIONS:
Overall Officials: I-Te Lee, Principal Investigator — Taichung Veterans General Hospital
Locations (1):
- Taichung Veterans General Hospital, Taichung, Taiwan

IPD SHARING:
Plan to Share IPD: No